CLINICAL TRIAL: NCT00379665
Title: Intratumoral Cancer Chemotherapy Through a Flexible Bronchoscope as an Adjunct to Brachytherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCT 05-01
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung; Chemotherapy; Cisplatin; Intratumoral; Bronchoscope; Brachytherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin (Experimental): 1 mg/ml at a dosage of approximately 2 mg per cubic cm of tumor. Weekly up to 6 injections.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — 1 mg/ml at a dosage of approximately 2 mg per cubic cm of tumor. Weekly up to 6 injections.

SUMMARY:
This study is being conducted in order to determine if intratumoral chemotherapy will be helpful in the palliation of endobronchial tumors when used in conjunction with endobronchial brachytherapy.

DETAILED DESCRIPTION:
Injections of cisplatin are given in conjunction with the brachytherapy procedure. If the direct intratumoral injections result in a decrease in the endobronchial obstructed airways and if the therapy is well tolerated, there will be immediate clinical benefit to this minimally invasive method, the most obvious being an improved quality of life. Approximately 2 mg cisplatin per cubic centimeter of tumor are injected into each tumor through a flexible bronchoscope. A total of four to six injections are administered one week apart. Response to therapy is assessed based on improvement in intraluminal obstruction by tumor, as assessed by endobronchial observation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable lung carcinoma and/or recurrent disease.
* Patients with symptomatic obstruction.
* Occlusion or partial occlusion of bronchi.
* Disease verified via bronchoscopy.
* Patients with a least one endobronchial tumor, measuring at least 0.5 cm.
* Patients between ages of 20 and 80 years.
* Documented informed consent must be obtained.

Exclusion Criteria:

* Patients without diagnosis confirmed by bronchoscopy.
* Patients with endobronchial tumors measuring less than 0.5 cm.
* Patients younger than 20 or older than 80 years.
* Patients who do not sign informed consent form.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-10; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To affect a faster clearing of the obstruction as compared with initial evaluation, based on the percentage of lumen opened. | within 4 to 6 injections

SECONDARY OUTCOMES:
Respiratory symptoms due to occlusion to be assessed both before and after the procedure. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nader, DO, Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center, Inc.
Locations (1):
- Cancer Treatment Centers of America ® Southwestern Regional Medical Center, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] BATEMAN JC. Palliation of cancer in human patients by maintenance therapy with NN'N"-triethylene thiophosphoramide and N-(3-oxapentamethylene)-N'N"-diethylene phosphoramide. Ann N Y Acad Sci. 1958 Apr 24;68(3):1057-71. doi: 10.1111/j.1749-6632.1958.tb42664.x. No abstract available. PMID 13627755
- [Background] Burris HA 3rd, Vogel CL, Castro D, Mishra L, Schwarz M, Spencer S, Oakes DD, Korey A, Orenberg EK. Intratumoral cisplatin/epinephrine-injectable gel as a palliative treatment for accessible solid tumors: a multicenter pilot study. Otolaryngol Head Neck Surg. 1998 Apr;118(4):496-503. doi: 10.1177/019459989811800412. PMID 9560102
- [Background] Monga SP, Wadleigh R, Adib H, Harmon JW, Berlin M, Mishra L. Endoscopic treatment of gastric cancer with intratumoral cisplatin/epinephrine injectable gel: a case report. Gastrointest Endosc. 1998 Oct;48(4):415-7. doi: 10.1016/s0016-5107(98)70014-8. No abstract available. PMID 9786117
- [Background] Vogl TJ, Engelmann K, Mack MG, Straub R, Zangos S, Eichler K, Hochmuth K, Orenberg E. CT-guided intratumoural administration of cisplatin/epinephrine gel for treatment of malignant liver tumours. Br J Cancer. 2002 Feb 12;86(4):524-9. doi: 10.1038/sj.bjc.6600116. PMID 11870531
- [Background] Celikoglu F, Celikoglu SI. Intratumoural chemotherapy with 5-fluorouracil for palliation of bronchial cancer in patients with severe airway obstruction. J Pharm Pharmacol. 2003 Oct;55(10):1441-8. doi: 10.1211/0022357021936. PMID 14607028
- [Background] Celikoglu SI, Celikoglu F, Goldberg EP. Intratumoral cancer chemotherapy through a flexible bronchoscope. J Bronchol. 2004;11:260-265.
- [Background] Goldberg EP, Hadba AR, Almond BA, Marotta JS. Intratumoral cancer chemotherapy and immunotherapy: opportunities for nonsystemic preoperative drug delivery. J Pharm Pharmacol. 2002 Feb;54(2):159-80. doi: 10.1211/0022357021778268. PMID 11848280